CLINICAL TRIAL: NCT01367054
Title: Adverse Events in Pharmaceutical Bioequivalence Study of Two Formulations of Metformine Hydrochloride 500 mg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocinese (Industry)
Responsible Party: Josélia Larger Manfio, Biocinese
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 06/2008; Met 2005 (Other: Biocinese)
Record Dates: First submitted 2011-04-27; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-05

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: Metformine; adverse events; bioequivalence
MeSH Terms: conditions — Nutritional and Metabolic Diseases | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): 500 mg
  Interventions: Drug: Metformin; Drug: Glifage

INTERVENTIONS:
Drug: Metformin — 500 mg tablet
  Other Names: Test
Drug: Glifage — 500 mg tablet
  Other Names: Reference

SUMMARY:
The objective is evaluate, in healthy volunteers, the bioavailability of two products containing metformine 500 mg to determine if they are bioequivalent and identify the occurrence of adverse events.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate, in healthy volunteers, the bioavailability of two products containing metformine 500 mg to determine if they are bioequivalent and identify the occurrence of adverse events.

MATERIAL AND METHODS: The study was approved by research Ethics Committee and all twenty-eight volunteers signed the selected IC. An open, randomized, crossover study with two periods of confinement and an interval of seven days between them was performed. Twenty (20) blood collections were performed between 30 minutes and 36 hours after drug administration. Plasma samples were analyzed by liquid chromatography mass spectrometry (LC-MS/MS). Statistical analysis was conducted based on pharmacokinetic parameters: maximum concentration (Cmax) and area under the curve (AUC 0-te AUC 0-inf). Analysis of variance (ANOVA) model appropriate was employed for the two periods cross under the logarithmically transformed data.

ELIGIBILITY:
Inclusion Criteria:

* Within 10% of their ideal body weight
* Age between 18 and 50 years
* Healthy conditions
* Ability to understand the written informed consent

Exclusion Criteria:

* Pregnancy
* Smokers
* Alcohol and drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Participants will be followed for the duration of hospital stay, an expected average of 24 hours. All adverse events observed are analyzed.
  Observation of adverse events after a single dose. After administration, the volunteers need to answer the question: how are you? All complains are registered. The adverse events are going to be classified as linked ou not with the drug. The expected result is "x" volunteers presented adverse events, the most frequent was "y" event, and so one.

CONTACTS AND LOCATIONS:
Overall Officials: Josélia Manfio, Dr, Principal Investigator — Biocinese
Locations (1):
- Biocinese, Toledo, Paraná, Brazil